CLINICAL TRIAL: NCT02719301
Title: Necklace-Shaped Sensor for Non-Invasive Monitoring of Stroke Volume, Cardiac Output, Fluids, Heart Rate, Heart Rate Variability, and Respiration Rate
Brief Title: Necklace-Shaped Sensor for Non-Invasive Monitoring of Stroke Volume and Cardiac Output
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PERM-IRB-001-CM
Record Dates: First submitted 2016-03-17; First posted 2016-03-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men/Women between 18 & 85: Accepting both healthy and non-healthy subjects. A portion of the subjects will have a fluid management issue or heart failure.

SUMMARY:
Study will compare measurements made with Necklace device for stroke volume/cardiac output with values from a FDA-approved reference device. The gold standard that will be used is Cardiac MRI. Subjects will be measured with both the Necklace, reference device, and the Cardiac MRI. Values calculated by the Cardiac MRI analysis will be compared with the reference device and the Necklace.

DETAILED DESCRIPTION:
Study will compare measurements made with Necklace device for stroke volume/cardiac output with values from a FDA-approved reference device. The gold standard that will be used is Cardiac MRI. Subjects will be measured with both the Necklace, reference device, and the Cardiac MRI. Values calculated by the Cardiac MRI analysis will be compared with the reference device and the Necklace.

The Cardiac MRI will be received ~1-4 days after the measurement is completed. The data will be compared with data collected from the Necklace and the reference device during the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to undergo Cardiac MRI

Exclusion Criteria:

* Sensitivity to electrodes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and Women between 18 and 85.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Stroke Volume Measurement from Necklace with Cardiac MRI measurement of Stroke Volume | Retrospective up to 6 months after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Banet, Principal Investigator — Baxter Healthcare Corporation

IPD SHARING:
Plan to Share IPD: No